Committee of Scientific Research
Department of Athletic sciences
Decision number: UoM.S-1/24

Date: 02/June/2024



Ministry of Higher Education and Scientific Research University of Mosul College of Physical Education and Sport Sciences

## **Scientific Research Committee Decision**

The scientific research committee for Athletic Sciences Department of College of Physical Education and Sport Sciences at University of Mosul has discussed the research protocol number UoM-S1/24 which is entitled:

(Feasibility a combining rehabilitation program at field exercises and tele-exercises to enhance daily life activities to rural women in Iraq)

Submitted by researchers:

(Munib Abdullah Fathe, Amal Machfer, Stevan Karash, Mohamed Amine Bouzid, Hamdi Chtourou, and Wassim Moalla)

To the scientific research committee to obtain the ethical approval, the committee has decided to accept the above-mentioned research protocol as it meets the standard adopted by Ministry of Higher Education and Scientific Research, University of Mosul, College of Physical Education and Sport Sciences, and in strict accordance with recognized scientific and ethical principles, including those outlined in the Declaration of Helsinki, and there is no objection to implementing it this field. Please be advised that this approval is valid from the date of this letter until the study's end date as indicated in your application. If you plan to extend the study period or make any significant changes to the research protocol, you must notify the committee in advance by submitting an amendment request.



## Notes:

- -The Committee Chairperson/Committee aperture was authorized to sign this decision on behalf of the remaining members of the committee under the rules of procedure of the scientific research committee
- The approval means that the research project submitted to the aforementioned committee has fulfilled the ethical and methodology standard adopted by University of Mosul.